CLINICAL TRIAL: NCT03382691
Title: M- HEALTHCARE Confirmatory Clinical Trials Used for Measurement of the ABP for the Accuracy and Safety Assessment of the Module Measuring Blood Pressure
Brief Title: Accuracy of a Blood Pressure Measuring Mobile Device in Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Seoul National University Bundang Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SNUBH_GO_056
Record Dates: First submitted 2017-10-29; First posted 2017-12-26 (Actual); Last update posted 2017-12-26 (Actual); Status verified 2017-10

CONDITIONS: Blood Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXPERIMENTAL (Experimental): Blood pressure check using mobile device and control device
  Interventions: Device: blood pressure check

INTERVENTIONS:
Device: blood pressure check — Check blood pressure using new device and conventional device alternatively. Compare blood pressure measured with new device and conventional device.

SUMMARY:
The accuracy and safety of blood pressure module of new mobile device (M- HEALTHCARE device) is evaluated according to Korean FDA guidelines in 100 healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Participants whose systolic blood pressure <=110 should be at least 10% of whole cohort
2. Participants whose systolic blood pressure >=160 should be at least 10% of whole cohort
3. Participants whose diastolic blood pressure >=100 should be at least 10% of whole cohort
4. Participants whose diastolic blood pressure <=70 should be at least 10% of whole cohort
5. Participants whose arm circumference are between 20cm and 30cm should be 25 - 50% of whole cohort
6. Participants whose arm circumference are between 30cm and 40cm should be 50 - 75% of whole cohort

Exclusion Criteria:

1. heart disease with abnormal rhythm
2. peripheral vascular anomaly or disease
3. inadequate to be applied blood pressure cuff (e.g. trauma on arm)
4. pregnant or lactating women

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
mean difference of systolic blood pressure | 1 day at visit 2
  mean difference of blood pressure between new and control device
mean difference of diastolic blood pressure | 1 day at visit 2
  mean difference of diastolic blood pressure between new and control device
standard deviation of the difference of systolic blood pressure | 1 day at visit 2
  standard deviation of the difference of systolic blood pressure between new and control device
standard deviation of the difference of diastolic blood pressure | 1 day at visit 2
  standard deviation of the difference of diastolic blood pressure between new and control device

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyenggi DO, South Korea

IPD SHARING:
Plan to Share IPD: No